CLINICAL TRIAL: NCT01138527
Title: Prostate Cancer Localization With a Multiparametric MR Approach
Brief Title: Prostate Cancer Localization With a Multiparametric Magnetic Resonance (MR) Approach
Acronym: PCa-MAP
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Siemens AG (Industry); Mount Vernon Hospital (Other); Multi-Imagem and CDPI, Rio de Janeiro, Brasil (Unknown); Norwegian University of Science and Technology (Other); University of California, Los Angeles (Other); University Hospital, Ghent (Other); Johns Hopkins University (Other); Medical University of Vienna (Other); University Health Network, Toronto (Other); Heidelberg University (Other)
Responsible Party: Sponsor
Other Study IDs: RU PCa-MAP
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
Keywords: multi-parametric MRI approach
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fixed histopathology slides of resected prostates at local institutions: Not different from clinical routine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biopsy-proven prostate cancer: Patients with biopsy-proven prostate cancer, planned for radical prostatectomy
  Interventions: Other: MRI examination

INTERVENTIONS:
Other: MRI examination — 45-minute MRI examination of the prostate and surrounding tissues with T2-weighted MRI, diffusion-weighted MRI, Spectroscopic Imaging and dynamic contrast enhanced imaging

SUMMARY:
The primary objective of this prospective multi-centre study is to prove the diagnostic accuracy of in vivo 3T multi-modality Magnetic Resonance Imaging (high resolution T2-weighted MRI, DCE-MRI, MRSI and DWI techniques) in distinguishing carcinoma from other prostate tissue. The gold standard for distinguishing the tissue types is the analysis of whole-mount sections of the resected prostate by a genitourinary histopathologist.

DETAILED DESCRIPTION:
Goal Proving that multi-parametric MR imaging in a multi-centre setting allows for localizing clinically significant (volume > 0.5cc; Gleason > 6) prostate carcinoma in the prostate.

Objective 1

To determine the diagnostic accuracy (area under the receiver-operating characteristic curve) of 3-Tesla multi-modality non-endorectal coil (ERC) MR imaging in localizing prostate cancer, by correlating:

1. focal areas of low signal intensity on T2-weighted images;
2. the extent and degree of deviating metabolite ratios derived from MRSI. This can be the choline+creatine/citrate ratio or if possible, the choline / citrate ratio;
3. the extent and degree of apparent diffusion coefficient reduction on DWI;
4. the extent and degree of perfusion abnormality on DCE-MRI; with the presence or absence of cancer at (reconstructed) whole mount section histopathology.

Objective 2 Proving that multi-modality MR data allows for predicting tumor grade. The parameters from the different MR methods for a tumor focus can be correlated to the local Gleason grade of the corresponding lesion in the histopathological specimens.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diagnosis of adenocarcinoma of the prostate
* Subject will sign a consent form prior to study entry
* Radical prostatectomy and histopathological exam planned
* The time interval between last biopsy and the MR exam must be at least 4 weeks
* The time interval between MR exam and radical prostatectomy should not exceed 12 weeks

Exclusion Criteria:

* Subjects who are unable to give valid informed consent
* Subjects who are unwilling or unable to undergo an MR exam, including subjects with contra-indications to MR exams
* Therapy or surgical procedure applied to the prostate or to other organs in vicinity to the prostate: among the therapies preventing inclusion are any form of radiation therapy, cryo-therapy, thermal-therapy, therapy based on any other medication (including hormonal therapy).
* Patients under hormone deprivation therapy.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Biopsy-proven patients with prostate cancer, planned for radical prostatectomy.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2010-06; Primary Completion 2015-08 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Area under the ROC curve to distinguish between cancer and non-cancer tissue in the prostate | December 2015

SECONDARY OUTCOMES:
Area under the ROC curve to separate low aggressive from intermediate and high aggressive prostate cancer | december 2015

CONTACTS AND LOCATIONS:
Overall Officials: Tom W Scheenen, PhD, Principal Investigator — Radiology, Radboud University Nijmegen Medical Centre; Jurgen J Fütterer, MD PhD, Principal Investigator — Radiology, Radboud University Nijmegen Medical Centre
Locations (9):
- United States (2):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
- Medical University Vienna, Vienna, Austria
- Ghent University Hospita, Ghent, Belgium
- University Health Network, Princess Margaret Hospital, Toronto, Canada
- University Medical Center Mannheim, Heidelberg University, Mannheim, Germany
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands
- Norwegian University of Science and Technology, Trondheim, Norway
- Mount Vernon Hospital, Paul Strickland Scanner Centre, London, United Kingdom